CLINICAL TRIAL: NCT03917511
Title: Effects of Combined Robot-assisted Therapy With Mirror Priming on Hand Function and Health-related Conditions in Patients With Stroke.
Brief Title: Effects of Combined Robot-assisted Therapy With Mirror Priming in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201801025B0
Record Dates: First submitted 2019-01-08; First posted 2019-04-17 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-06

CONDITIONS: Chronic Stroke
Keywords: Stroke; Mirror therapy; Robotic Training; Neurorehabilitation
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic training with mirror therapy (Experimental): 20 minutes mirror therapy followed by 40 minutes robotic-assisted training
  Interventions: Behavioral: Robotic training with mirror therapy
- Robotic-assisted training (Sham Comparator): 20 minutes sham mirror therapy followed by 40 minutes robotic-assisted training
  Interventions: Behavioral: Robotic-assisted training

INTERVENTIONS:
Behavioral: Robotic training with mirror therapy — Participants will receive 18 intervention sessions for about 6 consecutive weeks in a clinical setting (1 hour per session, 3 sessions per week). For each intervention session, participants will first receive 20 minutes mirror therapy followed by 40 minutes robotic-assisted training (robotic-assisted training includes 10 minutes active/passive training mode and 30 minutes robot-participant interactive training mode).
  Arms: Robotic training with mirror therapy
Behavioral: Robotic-assisted training — The training procedure will be the same as the robotic-assisted training with mirror therapy group except that sham mirror therapy will be provided in the first 20 minutes in the intervention session.
  Arms: Robotic-assisted training

SUMMARY:
The purpose of this study is to examine the effects of combining robotic-assisted training and mirror therapy on upper extremity motor and physiological function, daily functions, quality of life and self-efficacy in stroke patients.

DETAILED DESCRIPTION:
Based on trigger theory, this study designed a combining robotic-assisted training and mirror therapy. Before robotic-assisted training, a mirror therapy is performed to double the healing effect of robotic-assisted training.

This study hypothesized that combining robotic-assisted training and mirror therapy can improve the performance of hand function in stroke patients and promote daily life function, quality of life, and self-efficacy compared to single machine-assisted therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Brain injury more than 3 months.
2. Modified Ashworth Scale proximal part ≤ 3, Modified Ashworth Scale distal part ≤ 2, and no serious muscle spasms.
3. The myoelectric signal can be detected to activate the instrument
4. unilateral paresis (FMA score<60)
5. no serious cognitive impairment (i.e., Mini Mental State Exam score > 24)
6. can provide informed consent

Exclusion Criteria:

1. Other neurological disease
2. Complete sense of body defect
3. Inability to understand instructions
4. current participation in any other research
5. Botulinum Toxin injection within 3 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Change scores of Fugl-Myer Assessment (FMA) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The UE-FMA subscale will be used to assess the sensorimotor impairment level of UE in patients after stroke. The UE-FMA contains 33 movements with a score range from 0 to 66. A higher UE-FMA score indicates less impairment of the paretic limb. The validity and reliability of FMA is good to excellent.
Change scores of Active Range of Motion (AROM) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  Patient performs the exercise to move the joint without any assistance to the muscles surrounding the joint.
Change scores of grip and pinch power(Jamar hand dynamometer) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Jamar hand dynamometer is the most widely cited in the literature and accepted as the gold standard by which other dynamometers are evaluated. Excellent concurrent validity of the Jamar hand dynamometer is reported. The Jamar hand dynamometer measure the grip-strength. The norm of healthy male aged 18 to 75 years is from 64.8 lb to 121.8 lb, while the norm of healthy female aged 18 to 75 years is from 41.5 lb to 78.7 lb. Higher value represent a greater grip-strength.
Change scores of MyotonPro | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  Investigators will use the MyotonPRO device to evaluate the viscoelastic properties of UE muscles.
Change scores of Modified Ashworth Scale (MAS) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The MAS is a 6-point ordinal scale that measures muscle spasticity in patients with brain lesions. Higher score indicates higher muscle tone. Investigators will assess the MAS scores of UE muscles, including biceps, triceps, wrist flexors and extensors, and finger flexors and extensors. The validity and reliability of MAS for patients with stroke were established to be adequate to good.
Change scores of Medical Research Council scale (MRC) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The MRC is an ordinal scale that assesses muscle strength. The scoring for each muscle ranges from 0 to 5, with a higher score indicates stronger muscle. The reliability of MRC for all muscle groups was good to excellent in patients with stroke.
Change scores of pressure pain threshold | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Commander Algometer (JTECH Medical, USA) is designed for easy handling and fine resolution to identify clinically significant pain sensitivity changes. The Commander Algometer provides a convenient, efficient, objective pain evaluation tool for treatment planning, progress evaluation and case management. The measured pressure thresholds/tolerances and trigger point tenderness will be reported by patients.
Change scores of Revised Nottingham Sensory Assessment (RNSA) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  Changes in sensation before and after intervention will be measured with rNSA. Tactile sensation,proprioception, and stereognosis will be assessed with various sensory modalities. The rNSA is scored based on a 3-point ordinal scale (0-2) with a higher score indicates better sensation. The psychometric properties of rNSA have been established in patients with stroke.
Change scores of Wolf Motor Function Test (WMFT) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Wolf Motor Function Test evaluates upper extremity motor function via 15 function-based tasks and 2 strength-based tasks. The Wolf Motor Function Test -time evaluates the time required to complete the function-based tasks, and the Wolf Motor Function Test -quality assesses functional ability on a 6-point ordinal scale. A lower Wolf Motor Function Test -time performance indicates faster movement, whereas a higher Wolf Motor Function Test -quality score suggests better quality of movement. The psychometric properties of Wolf Motor Function Test have been established in stroke patients.
Change scores of Jamar hand dynamometer | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Jamar hand dynamometer is the most widely cited in the literature and accepted as the gold standard by which other dynamometers are evaluated. Excellent concurrent validity of the Jamar hand dynamometer is reported. The Jamar hand dynamometer measure the grip-strength. The norm of healthy male aged 18 to 75 years is from 64.8 lb to 121.8 lb, while the norm of healthy female aged 18 to 75 years is from 41.5 lb to 78.7 lb. Higher value represent a greater grip-strength.
Change scores of Mini-Mental State Exam (MMSE) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Mini-Mental State Examination (MMSE) is the most commonly administered psychometric screening assessment of cognitive functioning. The MMSE is used to screen patients for cognitive impairment, track changes in cognitive functioning over time, and often to assess the effects of therapeutic agents on cognitive function. The total score of MMSE ranged from 0 to 30. Higher values represent a better cognitive functioning.
Change scores of Motor Activity Log (MAL) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Motor Activity Log evaluates the amount of use (AOU) and quality of movement (QOM) of the affected hand in completing 30 common daily tasks. Scoring of each task ranges from 0 to 5, with higher scores indicating more use or better movement quality. The responsiveness, validity, and reliability have been established in stroke patients.
Change scores of Nottingham Extended Activities of Daily Living Scale (NEADL) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The NEADL is a self-report scale that measures instrumental activities of daily living. It evaluates 4 areas of daily living, including mobility, kitchen, domestic, and leisure activities. The total score is 0-66, and a higher score indicates better daily functional ability. The psychometric properties of NEADL have been well established.
Change scores of Stroke Impact Scale (SIS) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The SIS 3.0 will be used to evaluate health-related quality of life for patients with stroke. The SIS assesses eight domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, and participation/role function) with 59 test items.
Change scores of stroke self-efficacy questionnaire (SSEQ) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  the Stroke Self-Efficacy Questionnaire (SSEQ) , a questionnaire developed to measure the most relevant self-efficacy and self-management domains specific to the stroke population. It contains 13 items that are rated on a 0 - 10 scale, with higher scores indicating greater levels of self-efficacy. Questionnaire includes a range of relevant functional tasks such as walking, getting comfortable in bed, as well as some self-management tasks.
Change scores of Daily Living Self-Efficacy Scale (DLSES) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The DLSES is designed to measure self-efficacy in psychosocial functioning and self-efficacy in activities of daily living, regardless of level of physical impairment.
Change scores of Functional Abilities Confidence Scale (FACS) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Functional Abilities Confidence Scale (FACS) was designed to measure the degree of self-efficacy or confidence a patient exhibits with various movements or postures.

SECONDARY OUTCOMES:
Kinematic Analysis | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline)
  The movements of the arm and trunk will be captured by a 7-camera motion analysis system during unilateral and bilateral reaching tasks. Kinematic variables, such as reaction time, movement time, peak velocity, path length during the tasks can assess a patient's motor function in daily activities after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

REFERENCES:
- [Derived] Chen YW, Li KY, Lin CH, Hung PH, Lai HT, Wu CY. The effect of sequential combination of mirror therapy and robot-assisted therapy on motor function, daily function, and self-efficacy after stroke. Sci Rep. 2023 Oct 6;13(1):16841. doi: 10.1038/s41598-023-43981-3. PMID 37803096